CLINICAL TRIAL: NCT00619645
Title: Reduced Intensity Stem Cell Transplantation (RIST) for Patients With Hematological Malignancies Conditioned With Fludarabine and Busulfan
Brief Title: Donor Peripheral Stem Cell Transplant, Fludarabine, and Busulfan in Treating Patients With Hematologic Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC#196; 288263 (Other: UC Davis); UCD-196 (Other: UCDCC)
Record Dates: First submitted 2008-02-20; First posted 2008-02-21 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: recurrent adult acute myeloid leukemia; adult acute lymphoblastic leukemia in remission; refractory anemia with excess blasts; refractory anemia with ringed sideroblasts; refractory anemia; refractory cytopenia with multilineage dysplasia; previously treated myelodysplastic syndromes; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); chronic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; recurrent adult Hodgkin lymphoma; refractory multiple myeloma; recurrent adult acute lymphoblastic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; secondary acute myeloid leukemia; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; recurrent adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; recurrent adult Burkitt lymphoma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; de novo myelodysplastic syndromes; secondary myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts; Anemia, Refractory; Congenital Abnormalities; Leukemia, Myeloid, Chronic-Phase; Leukemia, Lymphocytic, Chronic, B-Cell; Hodgkin Disease; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma | interventions — Busulfan; Cyclosporine; fludarabine phosphate; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RIST for Heme malignancies (Other): Busulfan 3.3 mg/kg over 3 hours on day -6 and day -5 Fludarabine 30 mg/m2 IV over 30 minutes on day -6 to day -2 followed by Transplant followed by Immunosuppressive/GVHD therapy
  Interventions: Drug: busulfan; Drug: cyclosporine; Drug: fludarabine phosphate; Drug: mycophenolate mofetil; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Drug: busulfan
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: mycophenolate mofetil
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
Giving chemotherapy drugs, such as fludarabine and busulfan, before a donor peripheral stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil before and after the transplant may stop this from happening.

PURPOSE: This phase II trial is studying the side effects of giving donor peripheral stem cell transplant together with fludarabine and busulfan and to see how well it works in treating patients with hematologic cancers.

DETAILED DESCRIPTION:
OUTLINE:

* Conditioning regimen: Patients receive busulfan IV over 3 hours on days -6 and -5 and fludarabine phosphate IV over 30 minutes on days -6 to -2.
* Allogeneic peripheral blood stem cell transplant (PBSC): Patients undergo allogeneic PBSC on day 0.
* Immunosuppressive therapy/graft-versus-host disease (GVHD) prophylaxis: Patients achieve100% donor T-cell chimerism on day 30 without disease recurrence, and cyclosporine A (CSA) IV continuously over 24 hours or orally every 12 hours on days -1 to 60 followed by a taper until day 100 and oral mycophenolate mofetil (MMF) once every 12 hours on days 1-40, in the absence of ≥ grade 2 GVHD.

Patients with recurrent disease or < 100% donor T-cell chimerism (on day 30) undergo a 12-day CSA and MMF taper followed by escalating doses of previously collected donor leukocyte infusion every 4 weeks until 100% donor T-cell chimerism or disease regression, in the absence of ≥ grade 2 GVHD.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with any of the following:

  * Acute myeloid leukemia (AML), meeting 1 of the following criteria:

    * Recurrent disease in remission, defined as morphological remission with bone marrow aspirate/biopsy showing ≤ 5% within 4 weeks before the start of study treatment (cytogenetic or molecular remission is not required)
    * In first complete remission (CR1) with poor-risk cytogenetics, antecedent hematological disease (i.e., myelodysplasia), or treatment-related leukemia
  * Acute lymphoblastic leukemia (ALL), meeting 1 of the following criteria:

    * Recurrent disease in remission, defined as morphological remission with bone marrow aspirate/biopsy showing ≤ 5% within 4 weeks before the start of study treatment (cytogenetic or molecular remission is not required)
    * CR1 with Philadelphia chromosome or poor-risk cytogenetics
  * Chronic myelogenous leukemia (CML), meeting the following criteria:

    * First or second chronic phase

      * Must be documented disease progression after imatinib mesylate therapy OR documented lack of cytogenetic response 6 months post-imatinib mesylate initiation OR imatinib mesylate intolerance
  * Chronic lymphocytic leukemia (CLL), meeting the following criteria:

    * Recurrent disease after fludarabine-based therapy

      * Must have chemosensitive disease at the time of relapse, defined as greater than 50% reduction of WBC and lymphadenopathy
  * Recurrent Hodgkin lymphoma, recurrent non-Hodgkin lymphoma (NHL) (low-, intermediate-, or high-grade disease*), or transformed NHL, meeting 1 of the following criteria:

    * Received prior autologous transplantation and cytoreductive therapy at the time of relapse to achieve complete remission (CR) or CR/unconfirmed (CRu) as defined by the International Workshop
    * Relapsed disease that required more than 2 salvage regimens to achieve CR or CRu
  * Recurrent multiple myeloma, meeting the following criteria:

    * Must have received prior autologous transplantation and demonstrate chemosensitivity at the time of relapse, defined as greater than 50% reduction of M-component or plasma-cell marrow infiltration
  * Myelodysplastic syndrome

    * Refractory anemia (RA)/RA with ringed sideroblasts (RARS), refractory cytopenia with multilineage dysplasia (RCMD)/refractory cytopenia with multilineage dysplasia with ringed sideroblasts (RCMD-RS), or RA with excess blasts (RAEB) I, meeting the following criteria:

      * Must be transfusion-dependent and have an IPSS score ≥ 1.5, based on WHO criteria
      * No RAEB II or del(5q)
* No uncontrolled CNS metastases
* 5-6/6 HLA-matched sibling or 9-10/10 matched unrelated donor (both patient and donor) available

PATIENT CHARACTERISTICS:

* Karnofsky performance status ≥ 50%
* Serum creatinine ≤ 2 mg/dL
* Not pregnant
* Fertile patients must use effective contraception
* 50 years of age or older

  * Patients 18-50 years of age are eligible if meeting 1 of the following criteria:

    * Have a preexisting medical condition
    * Received prior therapy (i.e., autologous transplantation) and are considered to be too high risk for conventional myeloablative transplantation
* Must be willing to accept or comprehend irreversible sterility as a side effect of therapy
* No uncontrolled active infection
* No psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible
* Cardiac ejection fraction ≥ 30%
* Corrected pulmonary-diffusing capacity ≥ 35%
* No serologic evidence of infection with HIV
* No decompensated liver disease with serum bilirubin > 2.0 mg/dL

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-06; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol M. Richman, MD, Study Chair — University of California, Davis
Locations (1):
- University of California Davis Cancer Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- RIST for Heme Malignancies: Busulfan 3.3 mg/kg over 3 hours on day -6 and day -5 Fludarabine 30 mg/m2 IV over 30 minutes on day -6 to day -2 followed by Transplant followed by Immunosuppressive/GVHD therapy
  busulfan
  cyclosporine
  fludarabine phosphate
  mycophenolate mofetil
  allogeneic hematopoietic stem cell transplantation
  peripheral blood stem cell transplantation
Period: Overall Study
Arm/Group | RIST for Heme Malignancies
Started | 8
Completed | 7
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | RIST for Heme Malignancies
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 59.4 [53.7 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Day 100 Transplant-related Mortality
Description: Patients were followed for death and whether or not that death was attributed to the day 100 transplant via physician assessment for 24 months after day 100 transplant.
Time Frame: 24 months after day 100 transplant
Measure: Count of Participants; unit: Participants
Arm/Group | RIST for Heme Malignancies
Number analyzed (Participants) | 8
Participants | 1

2. Secondary Outcome: Number of Patients Without Progression After Day 100 Transplant
Description: All patients will be followed for progression for 24 months after their day 100 transplant.
Time Frame: 24 months after day 100 transplant
Population: This outcome was not collected/analyzed
Arm/Group | RIST for Heme Malignancies
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Patients Alive 24 Months Post Day 100 Transplant
Description: Patients will be followed for survival for 24 months post day 100 transplant.
Time Frame: 24 months post day 100 transplant
Measure: Count of Participants; unit: Participants
Arm/Group | RIST for Heme Malignancies
Number analyzed (Participants) | 8
Participants | 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected through Day 100 of treatment.
Arm/Group | RIST for Heme Malignancies
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RIST for Heme Malignancies (N=8)
Abdominal Pain (Gastrointestinal disorders) | 2
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 5
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4
Anorexia (Gastrointestinal disorders) | 2
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 5
blood bicarbonate decreased (Metabolism and nutrition disorders) | 1
constipation (Gastrointestinal disorders) | 1
cough (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine increased (Metabolism and nutrition disorders) | 2
Pruritic rash (Skin and subcutaneous tissue disorders) | 1
diarrhea (Gastrointestinal disorders) | 1
dizziness (Nervous system disorders) | 2
Duodenal hemorrhage (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Edema: head and neck (General disorders) | 1
Edema: trunk/genital (General disorders) | 1 — Left breast
esophageal pain (Gastrointestinal disorders) | 1
Eye disorder (Eye disorders) | 1
Fatigue (General disorders) | 7
Fatigue-lower mobility (General disorders) | 1
Fever (General disorders) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Gastritis (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 4
Hemoglobin (Blood and lymphatic system disorders) | 7
Hemorrhoids (Gastrointestinal disorders) | 1
Hyperbilirubinemia (Investigations) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypertension (Cardiac disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Insomnia (Psychiatric disorders) | 2
Leukocytes (Investigations) | 6
Leukopenia (Investigations) | 3
Lymphopenia (Investigations) | 6
Mucositis (Gastrointestinal disorders) | 1 — Small lesions
Mucositis (Gastrointestinal disorders) | 2
Muscle weakness (General disorders) | 1
Myalgia (General disorders) | 1
Myelitis (Nervous system disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Somnolence (Nervous system disorders) | 1
Neutrophil count decreased (Investigations) | 6
Oral hemorrhage (Gastrointestinal disorders) | 1
Pain-lower extremity (Musculoskeletal and connective tissue disorders) | 1
Petechia (General disorders) | 1
Platelet count decreased (Investigations) | 5
Rash NOS (Skin and subcutaneous tissue disorders) | 1
Rash desuamating (Skin and subcutaneous tissue disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Sweating (Skin and subcutaneous tissue disorders) | 1
Taste alteration (Gastrointestinal disorders) | 1
Tremor (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
weight loss (General disorders) | 1

LIMITATIONS AND CAVEATS:
This study was closed after only enrolling 8 patients and results were never published.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes